CLINICAL TRIAL: NCT05539638
Title: The Role of Circulating Tumour DNA in Head and Neck Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC21058
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma; Human Papillomavirus (HPV)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cancers of the throat, oropharyngeal squamous cell carcinoma (OPSCC), are highly prevalent across Scotland. Over the past 10 years, both global and Scottish cases of OPSCC have increased, particularly those associated with human papillomavirus (HPV). However there has been little change in techniques for diagnosis and monitoring. Although imaging technologies are improving, results of imaging are often indeterminate and clinicians require additional tools to make informed decisions. With this in mind our research team have established a range of blood- based tests which detect and monitor cancer DNA fragments shed by tumours into the blood stream in OPSCC patients. Our initial studies have shown that such tests, which are minimally invasive compared to surgical biopsy, hold the potential to provide an accurate, "real-time" method to monitor patient response to treatment, identify early relapse and assist in clinical decision making. The investigators aim to expand these results to assist clinical decisions for both virally associated and non-viral associated OPSCC. Following this, the investigators will focus on the poorest prognosis OPSCC group (non-HPV tumours) by applying state-of-the-art DNA detection and sequencing technologies to analyse tumour- derived DNA fragments in the bloodstream, to follow treatment response and to develop new methods for detecting relapse and resistance to treatment in OPSCC. Ultimately, the investigators envisage that the implementation of such genetic assays of tumours and the fragments that they release into the bloodstream will provide a transformative shift in the clinical assessment and quality of life of OPSCC patients in Scotland.

DETAILED DESCRIPTION:
Oropharyngeal squamous cell carcinoma (OPSCC) is an increasingly prevalent cancer type in Scotland, with an annual incidence rate of 23.4 per 100,000 of population in 2017 compared to 17.3 per 100,000 in 1993 [1]. This is due in part to an increased frequency of human papillomavirus (HPV) -related disease, which accounts for >70% of cases of OPSCC, and to continuing high rates of smoking. The current standard of care in OPSCC rests on clinical assessment and cross-sectional imaging followed by biopsy with histopathological diagnosis via immunohistochemistry (IHC) and PCR testing of the tumour for HPV. Follow-up is by chemo-radiotherapy (CRT) in most cases, with interval imaging to gauge post-treatment response to therapy and salvage surgery as required [2]. HPV+ve OPSCC has a generally good prognosis after treatment with CRT (3-year survival 82%), whilst HPV-ve OPSCC has a much poorer prognosis (3-year survival 57%)[3]. Surgical access to post-treatment OPSCC for biopsy can be difficult and even with recent advances in functional imaging there are still significant numbers of patients, at first presentation and at relapse, with indeterminate results [4]. The poor prognosis of HPV-ve disease and the major differences in prognosis and management between HPV+ve and -ve disease underline the importance of accurate identification of HPV status in patients with OPSCC and emphasise the need for more reliable markers of residual or recurrent disease.

The analysis of circulating tumour-derived DNA (ctDNA) from patient blood - "liquid biopsy" - represents a minimally invasive approach to cancer diagnosis and management, with the potential to transform clinical care through identification in blood ctDNA of actionable tumour-derived mutations, detection of minimal residual disease and early detection of disease recurrence [5]. There has been significant interest in developing liquid biopsy approaches in HPV+ve OPSCC, with several studies including our own indicating that real-time monitoring of HPV levels in plasma cell-free DNA (cfDNA) can accurately determine HPV status, indicate completeness of response to treatment and provide evidence of tumour recurrence earlier than routine surveillance and before symptomatic presentation [6-8] (Thomson et al 2020, MedRxiv). In HPV-ve OPSCC, a particular problem in Scotland due to high rates of smoking, no such blood-based markers are available. As well as the opportunities to validate and translate HPV cfDNA as a biomarker for remission and relapse in HPV+ve OPSCC, there is therefore a need to develop new diagnostic assays to assist clinical decision-making steps in the management of HPV-ve disease.

The investigators aim to carry out liquid biopsy studies that will improve diagnostic accuracy and clinical management of Scottish OPSCC patients. In HPV+ve OPSCC, The investigators will expand our existing cohort and prospectively evaluate the clinical utility of cfDNA HPV analysis as a biomarker for routine care. In HPV-ve patients, The investigators will study the development and evolution of HPV-ve disease through combined genomic analyses of tumour DNA and circulating cfDNA, with the aim of identifying blood-based biomarkers and new targets for personalised therapy in this poor prognosis form of OPSCC. Understanding the molecular events surrounding OPSCC development and responsiveness to treatment, and identifying biomarkers for blood-based disease monitoring stand to have a significant impact on patient survival and quality of life of Scottish patients with OPSCC. The work proposed here - built upon a strong foundation of pilot data and collaboration between academia and the NHS - will directly assist clinical care and treatment efficacy for OPSCC patients in Scotland.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oropharyngeal squamous cell carcinoma
* Both HPV positive and negative disease

Exclusion Criteria:

* Patients under 18 years of age
* Those who lack capacity to consent
* Patients with non-squamous cell carcinoma
* Patients with squamous cell carcinoma out with the oropharynx

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Number of participants/volunteers = 400 patients with oropharyngeal squamous cell carcinoma recruited over 3-4 sites then followed for a median of 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-08-14 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal monitoring of HPV+ve tumour burden through analysis of HPV cfDNA by ddPCR to assess treatment success and for early detection of relapse. | 3 years
  A sample of blood (approx. 20 ml) will be collected from each participant. Using ddPCR assays the blood samples will be analysed for the 5 most prevalent serotypes of HPV seen in OPSCC (HPV16, 18, 31, 33 & 35) allowing for the quantification of cfDNA present in the blood samples (HPV copies/ml). This will be repeated longitudinally at several time points to correlate HPV DNA levels (HPV copies/ml) with the standard of care (12 week post treatment imaging, salvage surgery and biopsy where indicated, and clinical follow up) and to formally measure assay predictive value.

SECONDARY OUTCOMES:
The determination of tumour burden in HPV-ve OPSCC biopsy's | 3 years
  The investigators aim to define the genomic aberrations present in each HPV-ve patient's tumour biopsy material by Whole Exome Sequencing (WES) of solid tumour biopsied or resected at presentation. Genomic DNA will be isolated from tumour DNA taken from tissue biopsy material using commercially available exome sequencing kits and DNA libraries prepared prior to sequencing at our local sequencing facility on an Illumina Nextseq, at a target coverage of 100X.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Tay, Principal Investigator — NHS Lothian; Catriona Douglas, Principal Investigator — NHS Greater Glasgow and Clyde; Robin Crosbie, Principal Investigator — NHS Lanarkshire; Jaiganesh Manickavasagam, Principal Investigator — NHS Tayside; Kim Ah-see, Principal Investigator — NHS Grampian
Locations (5):
- United Kingdom (5):
  - Ninewells Hospital, Dundee, DD2 1SG
  - Summerfield House - NHS Grampian, Aberdeen
  - Monklands Hospital ENT, Airdrie
  - The Royal Infirmiry, Edinburgh
  - Glasgow Royal Infirmary, Glasgow